CLINICAL TRIAL: NCT06912906
Title: Comparison of Two Strategies to Allow Mechanical Ventilation Separation Using Biphasic Airway Pressure Ventilation Without Any Synchronization (BIPAP) or Pressure Support Ventilation (PSV): a Randomized Feasibility Trial
Brief Title: Feasibility Study to Compare Two Ventilatory Modes for Mechanical Ventilation Weaning
Acronym: BIWEAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Piquilloud Imboden Lise, Attending Physician, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-00432
Record Dates: First submitted 2025-03-12; First posted 2025-04-06 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Mechanical Ventilation Weaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care: Pressure support ventilation (PSV) (No Intervention): Patient will be weaned from mechanical ventilation using the pressure support ventilation (PSV) modality accoring to the local standard of care.
- Biphasic positive airway pressure without any synchronisation (BIPAPasynchro) (Experimental): Patients will be managed with byphaisc positive pressure modality without any synchronisation (BIPAPasynchro) as soon as they are considered to be ready to initiate the weaning phase from mechanical ventilation. Lausanne adult intesive care physicians will be provided a protocol to help guide them with the setting of BIPAPasynchro, as this is different from standard clinical pratice.
  Interventions: Procedure: BIPAPasynchro: byphaisc positive pressure modality without any synchronisation

INTERVENTIONS:
Procedure: BIPAPasynchro: byphaisc positive pressure modality without any synchronisation — Patients will be switched to byphaisc positive pressure modality without any synchronisation (BIPAPasynchro) as soon as they are considered to be ready to initiate the weaning phase from mechanical ventilation. Lausanne adult intesive care physicians will be provided a protocol to help guide them with the setting of BIPAPasynchro, as this is different from standard clinical pratice.
  Arms: Biphasic positive airway pressure without any synchronisation (BIPAPasynchro)

SUMMARY:
We hypothesize that the ventilatory mode Bilevel Positive Airway Pressure without any synchronization (BIPAPasynchro) may facilitate the weaning process of patients intubated with acute hypoxiemic respiratory failure (AHRF) by obviating the problem of patient-ventilator asynchrony. In order to prove this hypothesis a large randomized controlled study should be perfromed comparing BIPAPasynchro versus pressure support ventilation (PSV), the most widely used ventilatory mode during the weaning process. In order to do so, a feasibility trial to demonstrate the ICU personnel can effectively use a non-standard ventilatory mode should be first performed. The objective of our study is, thus, to demonstrate the feasibility of using BIPAasynchro in the Lausanne Adult ICU.

DETAILED DESCRIPTION:
Bilevel Positive Airway Pressure without any synchronization (BIPAPasynchro) ventilation is a ventilatory modality that guarantees a minimal mandatory minute ventilation, even in deeply sedated patients, and allows free spontaneous breathing as soon as possible, without requiring synchronization between the patient and the ventilator. The hypothesis is that, as it obviates the problem of patient-ventilator asynchrony, it could reduce, compared to pressure support ventilation (PSV), the need of sedation, decrease diaphragmatic atrophy and accelerate the liberation from mechanical ventilation (weaning phase) without exposing the patients to further risks. Data seems to suggest a potential benefit of BIPAPasynchro over PSV, but no large randomized controlled trials have been performed to compare the two techniques; however, this cannot be done after first demonstrating that it is feasible to use BIPAPasynchro in the weaning process from mechanical ventilation in the intensive care unit.

The present project aims at assessing the feasibility of using a standardized BIPAP weaning strategy. It is thus a feasibility trial that assesses the adherence to the use of the mode. It is a randomized trial with two parallel groups in which we will compare the percentage of time effectively spent in the assigned mode, either BIPAP asynchro (intervention group) or PSV (control group), since the first switch from assist-control ventilation to assisted ventilation.

The study primary endpoint is the percentage of patients who spent at least 65% of the time (a priori-chosen cut-off) in the assigned mode (either BIPAPasynchro or PSV mode) since the first switch to assisted ventilation until successful liberation from mechanical ventilation. Liberation from mechanical ventilation (successful weaning) is defined as follows: 1) for intubated patients, we consider the patient weaned from ventilation when extubated without reintubation within 72 hours. 2) For tracheostomized patients, we consider the patient weaned from ventilation as soon as ventilated less than 12h over 24h during three consecutive days.

The secondary endpoints are divided in other-feasibility endpoints, safety endpoints and exploratory endpoints.

The study secondary feasibility endpoints are:

1. the proportions of participants who are switched to the non-assigned mode (cross-over from one study group to the other). Concretely, this refers to the situations where the patients in the PSV group are ventilated in BIPAPasynchro and the patients in the BIPAPasynchro group are ventilated in PSV.
2. The percentage of time spent in the non-assigned ventilatory mode since patient inclusion;
3. reasons for cross-over;
4. physicians refusal rate of patient enrolment;
5. reasons of physicians refusal if applicable;
6. recruitment rates.

   Secondary safety endpoints

   The study secondary safety endpoints are:
7. pneumothoraxes rate;
8. unplanned extubation rate;
9. rate of severe respiratory acidosis (pH < 7.20);
10. rate of severe respiratory alkalosis (pH > 7.55);
11. ventilation acquired pneumonia (VAP) rate (13).

    Secondary exploratory endpoints

    The study secondary exploratory endpoints are:
12. ventilator-free-days at day 28 from intubation (VFDs-28);
13. ventilator-free-days at day 28 from randomization;
14. duration of invasive mechanical ventilation between randomization and successful weaning, as defined in § 2.2.1;
15. duration of invasive mechanical ventilation between randomization and successful weaning, defined as no reintubation (or reventilation) during 7 days after extubation
16. number of tracheostomized patients during the weaning process;
17. number of patients matching the criteria for difficult or prolonged weaning (14).
18. length of ICU stay (censored at day 90 after randomization);
19. ICU-free days at day 90 from randomization;
20. length of Hospital stay (censored at day 90 from randomization);
21. hospital-free days at day 90 from randomization;
22. proportion of days with RASS less or equal -2 (for almost 50% of daily assessments) during invasive mechanical ventilation;
23. proportion of days with sedation during invasive mechanical ventilation;
24. proportion of days with neuromuscular blocking agents administration for ventilation facilitation during invasive mechanical ventilation;
25. ICU mortality (censored at day 90 from randomization);
26. hospital mortality (censored at day 90 from randomization).

This is a prospective, open-label, parallel-group, randomized feasibility trial taking place in the Adult ICU of the University Hospital of Lausanne, Switzerland. Due to the nature of the research, this is an open-label study. Patients will be randomized with a 1:1 ratio for receiving either BIPAPasynchro or PSV as soon as switching to assisted ventilation is considered as possible by the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Intubated ICU patient with acute respiratory failure;
* PaO2-FiO2 ratio of less than 300 mmHg (40 kPa) at least one hour after intubation;
* control or assist-control ventilation;
* expected duration of mechanical ventilation of more than 24 hours;
* clinician in charge considers that the patient can be switched to assisted ventilation (weaning phase start);
* informed consent obtained by the patient himself / legal representative or authorization received from independent physician

Exclusion Criteria:

* less than 18 years old;
* pregnant women (because of very different respiratory mechanics);
* severe obesity (BMI > 40 kg/m2);
* known obstructive pulmonary disease;
* expected death within one week or very poor prognosis with end-of-life care decision expected/treatment withdrawal;
* neurological disorders heavily influencing breathing pattern, like suspected or proven hypoxic brain injury, spinal injury above C8, severe traumatic brain injury, polyneuropathies (ex. Guillain-Barré, myasthenia gravis);
* home non-invasive ventilation prior to ICU admission, except CPAP for obstructive sleeping apnoea syndrome;
* tracheostomised at ICU admission;
* suspected or proven broncho-pleural fistulas;
* extracorporeal membrane oxygenation (ECMO) treatment;
* ICU admission for major burns;
* enrolment in other trial with competitive outcomes or treatment strategies;
* Known opposition to research participation if patient is not able to consent (eg patient with refused GC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of time spent in the mode of assisted ventilation assigned by the randomization | From enrollement until liberation from mechanical ventilation or date of death, whichever comes first, assessed up to 90 days

SECONDARY OUTCOMES:
The proportions of participants who are switched to the non-assigned mode (cross-over from one study group to the other) | From enrollement until liberation from mechanical ventilation or date of death, whichever comes first, assessed up to 90 days
  This refers to the situations where the patients in the PSV group are ventilated in BIPAPasynchro and the patients in the BIPAPasynchro group are ventilated in PSV.
The percentage of time spent in the non-assigned ventilatory mode since patient inclusion | From enrollement until liberation from mechanical ventilation or date of death, whichever comes first, assessed up to 90 days
Reasons for cross-over | From enrollement until liberation from mechanical ventilation or date of death, whichever comes first, assessed up to 90 days
  Reason why the patient is ventilated with another ventilatory mode compared to the one to which he was assigned at randomisation
Physicians refusal rate of patient enrolment | At time of potential enrollement
Reasons of physicians refusal if applicable | At time of potential enrollement
Recruitment rates | At time of enrollment
Pneumothoraxes rate | From enrollement until liberation from mechanical ventilation or date of death, whichever comes first, assessed up to 90 days
Unplanned extubation rate | From enrollement until liberation from mechanical ventilaton or death, whichever comes first, assessed up to 90 days
Rate of severe respiratory acidosis (pH < 7.20) | From enrollement until liberation from mechanical ventilation or date of death, whichever comes first, assessed up to 90 days
Rate of severe respiratory alkalosis (pH > 7.55) | From enrollement until liberation from mechanical ventilation or date of death, whichever comes first, assessed up to 90 days
Ventilation acquired pneumonia (VAP) rate | From enrollement until liberation from mechanical ventilation or date of death, whichever comes first, assessed up to 90 days
Ventilator-free-days at day 28 from intubation | from intubation to 28 days after intubation
Ventilator-free-days at day 28 from randomization | from randomization until 28 days after randomisation
Duration of invasive mechanical ventilation between randomization and successful weaning | from randomization until liberation from mechanical ventilation or death, whichever comes first, assessed up to 90 days
  Liberation from mechanical ventilation (successful weaning) is defined as follows: 1) for intubated patients, we consider the patient weaned from ventilation when extubated without reintubation within 72 hours. 2) For tracheostomized patients, we consider the patient weaned from ventilation as soon as ventilated less than 12h over 24h during three consecutive days.
Duration of invasive mechanical ventilation between randomization and successful weaning | from randomization until successful liberation from mechanical ventilation or death, whichever comes first, assessed up to up to 90 days
  Successful weaning defined as no reintubation (or reventilation) during 7 days after extubation
Number of tracheostomized patients during the weaning process | From enrollement until liberation from mechanical ventilaton or death, whichever comes first, assessed up to 90 days
Number of patients matching the criteria for difficult or prolonged weaning | From enrollement until liberation from mechanical ventilation or date of death, whichever comes first, assessed up to 90 days
  Difficult weaning defined as more than 1 day and less than 1 week and prolonged weaning defined as weaning duration of 1 week or more
Length of ICU stay | from randomization until 90 days after randomization
ICU-free days at day 90 from randomization | from randomization until 90 days after randomization
Length of Hospital stay | from randomization until 90 days after randomization
Hospital-free days at day 90 from randomization | from randomization until 90 days after randomization
Proportion of days with RASS less or equal -2 (for almost 50% of daily assessments) during invasive mechanical ventilation; | from first intubation until liberation from mechanical ventilation or death, whichever comes first, assessed up to 90 days
Proportion of days with sedation during invasive mechanical ventilation | from first intubation until liberation from mechanical ventilation or death, whichever comes first, assessed up to 90 days
Proportion of days with neuromuscular blocking agents administration for ventilation facilitation during invasive mechanical ventilation | from first intubation until liberation from mechanical ventilation or death, whichever comes first, assessed up to 90 days
ICU mortality | from randomization until 90 days after randomization
Hospital mortality | from randomization until 90 days after randomization

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Hospital of Lausanne, Lausanne, Canton of Vaud
  - Lausanne University Hospital (CHUV), Lausanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baum M, Benzer H, Putensen C, Koller W, Putz G. [Biphasic positive airway pressure (BIPAP)--a new form of augmented ventilation]. Anaesthesist. 1989 Sep;38(9):452-8. German. PMID 2686487
- [Background] Richard JM, Beloncle FM, Beduneau G, Mortaza S, Ehrmann S, Diehl JL, Prat G, Jaber S, Rahmani H, Reignier J, Boulain T, Yonis H, Richecoeur J, Thille AW, Declercq PL, Antok E, Carteaux G, Vielle B, Brochard L, Mercat A; REVA network. Pressure control plus spontaneous ventilation versus volume assist-control ventilation in acute respiratory distress syndrome. A randomised clinical trial. Intensive Care Med. 2024 Oct;50(10):1647-1656. doi: 10.1007/s00134-024-07612-3. Epub 2024 Sep 17. PMID 39287651
- [Background] Gama de Abreu M, Cuevas M, Spieth PM, Carvalho AR, Hietschold V, Stroszczynski C, Wiedemann B, Koch T, Pelosi P, Koch E. Regional lung aeration and ventilation during pressure support and biphasic positive airway pressure ventilation in experimental lung injury. Crit Care. 2010;14(2):R34. doi: 10.1186/cc8912. Epub 2010 Mar 16. PMID 20233399
- [Background] Richard JC, Lyazidi A, Akoumianaki E, Mortaza S, Cordioli RL, Lefebvre JC, Rey N, Piquilloud L, Sferrazza Papa GF, Mercat A, Brochard L. Potentially harmful effects of inspiratory synchronization during pressure preset ventilation. Intensive Care Med. 2013 Nov;39(11):2003-10. doi: 10.1007/s00134-013-3032-7. Epub 2013 Aug 9. PMID 23928898
- [Background] Katzenschlager S, Simon CM, Rehn P, Grilli M, Fiedler MO, Muller M, Weigand MA, Neetz B. Time-controlled adaptive ventilation in patients with ARDS-lack of protocol adherence: a systematic review. Crit Care. 2023 Feb 10;27(1):57. doi: 10.1186/s13054-023-04340-w. No abstract available. PMID 36765424
- [Background] Rathgeber J, Schorn B, Falk V, Kazmaier S, Spiegel T, Burchardi H. The influence of controlled mandatory ventilation (CMV), intermittent mandatory ventilation (IMV) and biphasic intermittent positive airway pressure (BIPAP) on duration of intubation and consumption of analgesics and sedatives. A prospective analysis in 596 patients following adult cardiac surgery. Eur J Anaesthesiol. 1997 Nov;14(6):576-82. doi: 10.1046/j.1365-2346.1994.00178.x. PMID 9466092
- [Background] Elrazek EA. Randomized prospective crossover study of biphasic intermittent positive airway pressure ventilation (BIPAP) versus pressure support ventilation (PSV) in surgical intensive care patients. Middle East J Anaesthesiol. 2004 Oct;17(6):1009-21. PMID 15651509
- [Background] Rose L, Hawkins M. Airway pressure release ventilation and biphasic positive airway pressure: a systematic review of definitional criteria. Intensive Care Med. 2008 Oct;34(10):1766-73. doi: 10.1007/s00134-008-1216-3. Epub 2008 Jul 17. PMID 18633595
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Jubran A, Grant BJ, Duffner LA, Collins EG, Lanuza DM, Hoffman LA, Tobin MJ. Effect of pressure support vs unassisted breathing through a tracheostomy collar on weaning duration in patients requiring prolonged mechanical ventilation: a randomized trial. JAMA. 2013 Feb 20;309(7):671-7. doi: 10.1001/jama.2013.159. PMID 23340588
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] Hadfield DJ, Rose L, Reid F, Cornelius V, Hart N, Finney C, Penhaligon B, Molai J, Harris C, Saha S, Noble H, Clarey E, Thompson L, Smith J, Johnson L, Hopkins PA, Rafferty GF. Neurally adjusted ventilatory assist versus pressure support ventilation: a randomized controlled feasibility trial performed in patients at risk of prolonged mechanical ventilation. Crit Care. 2020 May 14;24(1):220. doi: 10.1186/s13054-020-02923-5. PMID 32408883
- [Background] Roshdy A, Elsayed AS, Saleh AS. Airway Pressure Release Ventilation for Acute Respiratory Failure Due to Coronavirus Disease 2019: A Systematic Review and Meta-Analysis. J Intensive Care Med. 2023 Feb;38(2):160-168. doi: 10.1177/08850666221109779. Epub 2022 Jun 22. PMID 35733377
- [Background] Blanch L, Villagra A, Sales B, Montanya J, Lucangelo U, Lujan M, Garcia-Esquirol O, Chacon E, Estruga A, Oliva JC, Hernandez-Abadia A, Albaiceta GM, Fernandez-Mondejar E, Fernandez R, Lopez-Aguilar J, Villar J, Murias G, Kacmarek RM. Asynchronies during mechanical ventilation are associated with mortality. Intensive Care Med. 2015 Apr;41(4):633-41. doi: 10.1007/s00134-015-3692-6. Epub 2015 Feb 19. PMID 25693449
- [Background] Fredericks AS, Bunker MP, Gliga LA, Ebeling CG, Ringqvist JR, Heravi H, Manley J, Valladares J, Romito BT. Airway Pressure Release Ventilation: A Review of the Evidence, Theoretical Benefits, and Alternative Titration Strategies. Clin Med Insights Circ Respir Pulm Med. 2020 Feb 5;14:1179548420903297. doi: 10.1177/1179548420903297. eCollection 2020. PMID 32076372
- [Background] Yoshida T, Rinka H, Kaji A, Yoshimoto A, Arimoto H, Miyaichi T, Kan M. The impact of spontaneous ventilation on distribution of lung aeration in patients with acute respiratory distress syndrome: airway pressure release ventilation versus pressure support ventilation. Anesth Analg. 2009 Dec;109(6):1892-900. doi: 10.1213/ANE.0b013e3181bbd918. PMID 19923518
- [Background] Neumann P, Wrigge H, Zinserling J, Hinz J, Maripuu E, Andersson LG, Putensen C, Hedenstierna G. Spontaneous breathing affects the spatial ventilation and perfusion distribution during mechanical ventilatory support. Crit Care Med. 2005 May;33(5):1090-5. doi: 10.1097/01.ccm.0000163226.34868.0a. PMID 15891341
- [Background] Grassi A, Ferlicca D, Lupieri E, Calcinati S, Francesconi S, Sala V, Ormas V, Chiodaroli E, Abbruzzese C, Curto F, Sanna A, Zambon M, Fumagalli R, Foti G, Bellani G. Assisted mechanical ventilation promotes recovery of diaphragmatic thickness in critically ill patients: a prospective observational study. Crit Care. 2020 Mar 12;24(1):85. doi: 10.1186/s13054-020-2761-6. PMID 32164784
- [Background] Putensen C, Zech S, Wrigge H, Zinserling J, Stuber F, Von Spiegel T, Mutz N. Long-term effects of spontaneous breathing during ventilatory support in patients with acute lung injury. Am J Respir Crit Care Med. 2001 Jul 1;164(1):43-9. doi: 10.1164/ajrccm.164.1.2001078. PMID 11435237
- [Background] Downs JB, Douglas ME, Sanfelippo PM, Stanford W, Hodges MR. Ventilatory pattern, intrapleural pressure, and cardiac output. Anesth Analg. 1977 Jan-Feb;56(1):88-96. doi: 10.1213/00000539-197701000-00021. PMID 319705
- [Background] Saddy F, Moraes L, Santos CL, Oliveira GP, Cruz FF, Morales MM, Capelozzi VL, de Abreu MG, Garcia CS, Pelosi P, Rocco PR. Biphasic positive airway pressure minimizes biological impact on lung tissue in mild acute lung injury independent of etiology. Crit Care. 2013 Oct 8;17(5):R228. doi: 10.1186/cc13051. PMID 24103805
- [Background] Saddy F, Oliveira GP, Garcia CS, Nardelli LM, Rzezinski AF, Ornellas DS, Morales MM, Capelozzi VL, Pelosi P, Rocco PR. Assisted ventilation modes reduce the expression of lung inflammatory and fibrogenic mediators in a model of mild acute lung injury. Intensive Care Med. 2010 Aug;36(8):1417-26. doi: 10.1007/s00134-010-1808-6. Epub 2010 Mar 24. PMID 20333356